CLINICAL TRIAL: NCT06492824
Title: Intervention in Depression: Randomized Control Trial Examining a Fully Automated Mobile Behavioral Activation Intervention
Brief Title: Text Based Digital Interventions Prompting Enjoyable and Healthy Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Nick Santopetro, Co-Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003514
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Depression; Anhedonia
MeSH Terms: conditions — Depression; Anhedonia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enjoyable Activities Condition (Experimental): Watched an introduction video that discussed the rationale for the enjoyable activities intervention. During the initial visit, enjoyable activities participants were asked to choose five enjoyable activities from a large list that they wanted to do more frequently over the next four weeks. Over the next four weeks, daily text message reminders were sent each morning. These text messages reminded participants of the five enjoyable activities that they wanted to do and encouraged them to complete at least two of the of the enjoyable activities that day. Additionally, participants received a link to complete a daily checklist where they reported if they had completed any of their five activities on the previous day. At the end of the four-week period, enjoyable activities participants completed a post-intervention online survey consisting of the same measures from the initial survey.
  Interventions: Behavioral: Enjoyable Activities Condition
- Healthy Activities Condition (Active Comparator): Participants in the healthy activities condition were promoted to complete the following five activities each day: drinking more water, going to bed early, brushing their teeth, showering or bathing that day, and eating well-balanced meals. Healthy activities condition participants also watched an introduction video that discussed the rationale for the healthy activities intervention. Daily text reminders were sent regarding these five healthy living activities each morning. Consistent with the enjoyable activities condition, healthy activities participants were asked to try to complete at least two of the five healthy activities each day but could do more if they desired. At the end of the month, they completed an online post-intervention survey consisting of the same measures from the pre-intervention assessment.
  Interventions: Behavioral: Healthy Activities Condition
- Passive Control (No Intervention): Control participants completed an initial online survey which also included an introduction video (approximately one and half minutes long) explaining the rationale for this specific condition and that researchers wanted to understand the naturalistic course of mood and behavior over the course of one month. However, passive control participants were not explicitly asked to complete any enjoyable activities or healthy living activities during the subsequent four weeks. Passive control participants were not sent daily text reminders or checklists to complete over the four-week period. They were asked to complete the same short weekly questionnaire asking about their mood for the preceding week. At the end of the month, they also completed a post online survey consisting of the same measures from the initial survey. Participants in this condition also had the option to complete the enjoyable activities digital intervention after completing the passive control condition if they desired.

INTERVENTIONS:
Behavioral: Enjoyable Activities Condition — Participants complete an introduction video about the intervention. They will then take a pre-intervention survey, after which they will choose five enjoyable activities from a large list. Daily text message reminders will be sent to BA participants in the morning to remind them to do their enjoyable activities for the day, as well as a link to a checklist where they will report how frequently they have completed any of their five activities from the previous day (example text message in documentation). At the end of the month, they will complete a follow-up survey consisting of the same measures from the pre-intervention survey.
  Arms: Enjoyable Activities Condition
Behavioral: Healthy Activities Condition — They will take a pre-intervention survey and choose five enjoyable activities from the same list; however, active control participants will not explicitly be asked to complete these activities for the intervention. Participants in the active control condition will be promoted to complete tasks such as drinking more water, going to bed early, brushing their teeth, showering or bathing for that day, and eating well balanced meals. Daily text reminders will be sent about these healthy living activities in the morning. In that same message, they will receive a link to a checklist where they will report about their completed healthy living activities for the previous day (example text message in documentation). At the end of the month, they will also complete a follow-up survey consisting of the same measures from the pre-intervention survey.
  Arms: Healthy Activities Condition

SUMMARY:
The proposed project aims to examine the effectiveness of an automated digital (i.e., text message based) intervention prompting adults with at least moderate depressive symptoms to complete enjoyable daily activities (i.e., Behavioral Activation [BA]) over the course of one month compared to adults with moderate or more depressive symptoms that complete an active and a passive control condition broadly prompting a healthier lifestyle or no prompts at all. More specifically, we aim to examine if the BA intervention will improve mental health and overall well-being among adults experiencing moderate or more symptoms of depression over and beyond the active and passive control conditions. We will measure symptoms such as current depression, anxiety, and stress pre- and post- interventions to determine their effectiveness.

DETAILED DESCRIPTION:
Participants in the experimental (BA) condition will complete an introduction video about the intervention. They will then take a pre-intervention survey, after which they will choose five enjoyable activities from a large list. Daily text message reminders will be sent to BA participants in the morning to remind them to do their enjoyable activities for the day, as well as a link to a checklist where they will report how frequently they have completed any of their five activities from the previous day (example text message in documentation). At the end of the month, they will complete a follow-up survey consisting of the same measures from the pre-intervention survey.

Participants in the active control condition will complete mostly the same tasks as those in the experimental (BA) condition. They will then take a pre-intervention survey and choose five enjoyable activities from the same list; however, active control participants will not explicitly be asked to complete these activities for the intervention. Instead, participants in the active control condition will be promoted to complete tasks such as drinking more water, going to bed early, brushing their teeth, showering or bathing for that day, and eating well balanced meals. Daily text reminders will be sent about these healthy living activities in the morning. In that same message, they will receive a link to a checklist where they will report about their completed healthy living activities for the previous day (example text message in documentation).At the end of the month, they will also complete a follow-up survey consisting of the same measures from the pre-intervention survey. Importantly, participants in this condition will have the option to complete the BA digital intervention after completing the active control condition if they desire; however, these participants would not be paid for their time upon completing the BA intervention.

Finally, participants in the passive control condition will complete mostly the same tasks as those in the experimental (BA) and active control conditions. They will take a pre-intervention survey and choose five enjoyable activities from the same list; however, passive control participants will not explicitly be asked to complete these enjoyable activities or any of the healthy living activities during the month. To further clarify, passive control participants will not be enrolled in SlickText and will therefore not be sent daily text reminders or checklists. At the end of the month, they will also complete a follow-up survey consisting of the same measures from the pre-intervention survey. Importantly, participants in this condition will also have the option to complete the BA digital intervention after completing the passive control condition if they desire; however, these participants would not be paid for their time upon completing the BA intervention.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-8 score greater than or equal to 10
* 18 years or older
* Had access to a cell phone

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms | Collected at baseline and one month
  Depression, Anxiety, and Stress Scale (DASS-21) creates a total score for depression based on 7 items. Scores range from 0-42, higher score indication more depression.
Change in anhedonia | Collected at baseline and one month
  Personality Inventory for DSM-5 (PID 5), anhedonia subscale, creates a score of current anhedonic symptoms consisting of 8 items. Scores range from 0-24, higher scores indicating more symptoms of anhedonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT06492824/ICF_000.pdf